CLINICAL TRIAL: NCT06539234
Title: Angiotensin II Stress Test. Renin Kinetics During Treatment of Vasoplegic Shock With Angiotensin II in Relation to Hemodynamic Response to Treatment With Angiotensin II.
Brief Title: Angiotensin II Stress Test. Renin Kinetics During Treatment of Vasoplegic Shock With Angiotensin II.
Acronym: TENSINTEST
Status: Recruiting | Type: Observational
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Andreja Möller Petrun, MD, PhD, Assist. Prof. Andreja Möller Petrun, MD, PhD, University Medical Centre Maribor
Other Study IDs: UKC-MB-KME-33/24
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Shock; Vasoplegic Syndrome
Keywords: shock, distributive; angiotensin II; renin; shock, septic; vasoplegia
MeSH Terms: conditions — Shock; Vasoplegia; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Shock is a life-threatening condition which can cause multiple organ failure and even death. One characteristic of shock is low blood pressure which is managed with drugs called vasopressors. Most frequently used vasopressors are noradrenaline, vasopressin and recently also angiotensin II. Angiotensin II is present in the body and has a physiological role in maintaining blood pressure in healthy persons. Renin is an enzyme and a key factor in angiotensin II production in the body. In patients with shock, there is a lack of angiotensin II and an excess of renin in the body. Due to the literature renin has the potential to be a marker of severity of shock. Synthetic angiotensin II is used in patients with shock in whom we cannot normalize the blood pressure with noradrenaline and vasopressin. Regarding scientific data, the use of synthetic angiotensin II reduces the dose of noradrenaline and vasopressin and the incidence of acute kidney injury. The aim of our study is to find out what is the relation between the concentration of renin before and 6 hours after the start of using angiotensin II in patients with shock and their clinical outcome. Since not all patients with shock are responding to angiotensin II, the aim of our study is also to find out which patients could benefit most from synthetic angiotensin II.

DETAILED DESCRIPTION:
In patients with distributive shock (≥18 years) with noradrenaline >0,3 mcg/kg/min and vasopressin >0,03 IE/min not achieving an appropriate mean arterial pressure (65-85 mmHg) an angiotensin II infusion will be started at 20 ng/kg/min and after that adjusted to a max dose of 40 ng/kg/min if needed. Before the infusion and 6 hours after the start of angiotensin II infusion a blood sample will be drawn to determine the renin concentration. The primary outcome will be organ failure free days and ICU free days. Secondary outcome will be the need for vasopressors, dialysis, mechanical ventilation, trend of renin concentration.

ELIGIBILITY:
Inclusion Criteria:

* patients with distributive shock lasting < 72 hours
* a goal mean arterial pressure (65-85 mmHg) not achieved despite an infusion of at least noradrenaline 0.3 mcg/kg/min and vasopressin 0.03 IE/min
* the patient did not get angiotensin II before
* predicted survival is >24h
* no limitations for active treatment

Exclusion Criteria:

* burns >20% body area
* acute coronary syndrome
* bronchospasm
* liver disease (MELD ≥30)
* severe acute bleeding (need for 4 or more units of concentrated erythrocyte)
* acute mesenteric ischemia
* aortic dissection
* leucopenia <1000/mm3
* pregnancy
* Raynaud disease, systemic sclerosis, vasospastic disease
* the need for daily dose of hydrocortisone 500 mg or more
* ECMO

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (≥ 18 years old) with distributive shock (<72 hours duration) regardless of etiology without limitations for treatment and a predicted survival >24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
organ failure free days | 0-30 days
  days alive without the need of vasopressors, ventilators, or dialysis
ICU free days | 0-30 days
  30 minus the number of days in the ICU

SECONDARY OUTCOMES:
duration of the need for vasopressors | 0-30 days
  time in which vasopressors are needed
mechanical ventilation need | 0-30 days
  time of mechanical ventilation (invasive and/or noninvasive)
dyalisis need | 0-30 days
  time of eventual need for dyalisi´s
renin trend | 0-6 hours
  renin concentration before and 6 hours after the start of angiotensin II infusion

CONTACTS AND LOCATIONS:
Overall Officials: Andreja Möller Petrun, PhD, Study Chair — University Medical Centre Maribor
Locations (2):
- Slovenia (2):
  - Medical ICU, University Medical Centre Maribor, Maribor
  - Surgical ICU, University Medical Centre Maribor, Maribor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yehya N, Harhay MO, Curley MAQ, Schoenfeld DA, Reeder RW. Reappraisal of Ventilator-Free Days in Critical Care Research. Am J Respir Crit Care Med. 2019 Oct 1;200(7):828-836. doi: 10.1164/rccm.201810-2050CP. PMID 31034248
- [Background] Auriemma CL, Taylor SP, Harhay MO, Courtright KR, Halpern SD. Hospital-Free Days: A Pragmatic and Patient-centered Outcome for Trials among Critically and Seriously Ill Patients. Am J Respir Crit Care Med. 2021 Oct 15;204(8):902-909. doi: 10.1164/rccm.202104-1063PP. No abstract available. PMID 34319848
- [Background] De Backer D, Cecconi M, Chew MS, Hajjar L, Monnet X, Ospina-Tascon GA, Ostermann M, Pinsky MR, Vincent JL. A plea for personalization of the hemodynamic management of septic shock. Crit Care. 2022 Dec 1;26(1):372. doi: 10.1186/s13054-022-04255-y. PMID 36457089
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Vincent JL, Singer M, Einav S, Moreno R, Wendon J, Teboul JL, Bakker J, Hernandez G, Annane D, de Man AME, Monnet X, Ranieri VM, Hamzaoui O, Takala J, Juffermans N, Chiche JD, Myatra SN, De Backer D. Equilibrating SSC guidelines with individualized care. Crit Care. 2021 Nov 17;25(1):397. doi: 10.1186/s13054-021-03813-0. No abstract available. PMID 34789298
- [Background] Maslove DM, Tang B, Shankar-Hari M, Lawler PR, Angus DC, Baillie JK, Baron RM, Bauer M, Buchman TG, Calfee CS, Dos Santos CC, Giamarellos-Bourboulis EJ, Gordon AC, Kellum JA, Knight JC, Leligdowicz A, McAuley DF, McLean AS, Menon DK, Meyer NJ, Moldawer LL, Reddy K, Reilly JP, Russell JA, Sevransky JE, Seymour CW, Shapiro NI, Singer M, Summers C, Sweeney TE, Thompson BT, van der Poll T, Venkatesh B, Walley KR, Walsh TS, Ware LB, Wong HR, Zador ZE, Marshall JC. Redefining critical illness. Nat Med. 2022 Jun;28(6):1141-1148. doi: 10.1038/s41591-022-01843-x. Epub 2022 Jun 17. PMID 35715504
- [Background] Suzuki Y, Ruiz-Ortega M, Lorenzo O, Ruperez M, Esteban V, Egido J. Inflammation and angiotensin II. Int J Biochem Cell Biol. 2003 Jun;35(6):881-900. doi: 10.1016/s1357-2725(02)00271-6. PMID 12676174
- [Background] Laghlam D, Jozwiak M, Nguyen LS. Renin-Angiotensin-Aldosterone System and Immunomodulation: A State-of-the-Art Review. Cells. 2021 Jul 13;10(7):1767. doi: 10.3390/cells10071767. PMID 34359936
- [Background] Bitker L, Burrell LM. Classic and Nonclassic Renin-Angiotensin Systems in the Critically Ill. Crit Care Clin. 2019 Apr;35(2):213-227. doi: 10.1016/j.ccc.2018.11.002. Epub 2019 Jan 28. PMID 30784605
- [Background] Paul M, Poyan Mehr A, Kreutz R. Physiology of local renin-angiotensin systems. Physiol Rev. 2006 Jul;86(3):747-803. doi: 10.1152/physrev.00036.2005. PMID 16816138
- [Background] Correa TD, Takala J, Jakob SM. Angiotensin II in septic shock. Crit Care. 2015 Mar 16;19(1):98. doi: 10.1186/s13054-015-0802-3. PMID 25886853
- [Background] Garcia B, Zarbock A, Bellomo R, Legrand M. The alternative renin-angiotensin system in critically ill patients: pathophysiology and therapeutic implications. Crit Care. 2023 Nov 20;27(1):453. doi: 10.1186/s13054-023-04739-5. PMID 37986086
- [Background] Hall A, Busse LW, Ostermann M. Angiotensin in Critical Care. Crit Care. 2018 Mar 20;22(1):69. doi: 10.1186/s13054-018-1995-z. PMID 29558991
- [Background] Bellomo R, Zarbock A, Landoni G. Angiotensin II. Intensive Care Med. 2024 Feb;50(2):279-282. doi: 10.1007/s00134-023-07290-7. Epub 2024 Jan 8. No abstract available. PMID 38189932
- [Background] Forrester SJ, Booz GW, Sigmund CD, Coffman TM, Kawai T, Rizzo V, Scalia R, Eguchi S. Angiotensin II Signal Transduction: An Update on Mechanisms of Physiology and Pathophysiology. Physiol Rev. 2018 Jul 1;98(3):1627-1738. doi: 10.1152/physrev.00038.2017. PMID 29873596
- [Background] Sica DA. Angiotensin receptor blockers: new considerations in their mechanism of action. J Clin Hypertens (Greenwich). 2006 May;8(5):381-5. doi: 10.1111/j.1524-6175.2005.05141.x. PMID 16687949
- [Background] Busse LW, Barker N, Petersen C. Vasoplegic syndrome following cardiothoracic surgery-review of pathophysiology and update of treatment options. Crit Care. 2020 Feb 4;24(1):36. doi: 10.1186/s13054-020-2743-8. PMID 32019600
- [Background] Bronicki RA, Hall M. Cardiopulmonary Bypass-Induced Inflammatory Response: Pathophysiology and Treatment. Pediatr Crit Care Med. 2016 Aug;17(8 Suppl 1):S272-8. doi: 10.1097/PCC.0000000000000759. PMID 27490610
- [Background] Hall R. Identification of inflammatory mediators and their modulation by strategies for the management of the systemic inflammatory response during cardiac surgery. J Cardiothorac Vasc Anesth. 2013 Oct;27(5):983-1033. doi: 10.1053/j.jvca.2012.09.013. Epub 2012 Dec 29. No abstract available. PMID 23276596
- [Background] Paparella D, Yau TM, Young E. Cardiopulmonary bypass induced inflammation: pathophysiology and treatment. An update. Eur J Cardiothorac Surg. 2002 Feb;21(2):232-44. doi: 10.1016/s1010-7940(01)01099-5. PMID 11825729
- [Background] Levy B, Fritz C, Tahon E, Jacquot A, Auchet T, Kimmoun A. Vasoplegia treatments: the past, the present, and the future. Crit Care. 2018 Feb 27;22(1):52. doi: 10.1186/s13054-018-1967-3. PMID 29486781
- [Background] Squiccimarro E, Stasi A, Lorusso R, Paparella D. Narrative review of the systemic inflammatory reaction to cardiac surgery and cardiopulmonary bypass. Artif Organs. 2022 Apr;46(4):568-577. doi: 10.1111/aor.14171. Epub 2022 Jan 21. PMID 35061922
- [Background] Stoppe C, McDonald B, Benstoem C, Elke G, Meybohm P, Whitlock R, Fremes S, Fowler R, Lamarche Y, Jiang X, Day AG, Heyland DK. Evaluation of Persistent Organ Dysfunction Plus Death As a Novel Composite Outcome in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):30-8. doi: 10.1053/j.jvca.2015.07.035. Epub 2015 Jul 29. PMID 26847748
- [Background] Bernstein KE, Khan Z, Giani JF, Cao DY, Bernstein EA, Shen XZ. Angiotensin-converting enzyme in innate and adaptive immunity. Nat Rev Nephrol. 2018 May;14(5):325-336. doi: 10.1038/nrneph.2018.15. Epub 2018 Mar 26. PMID 29578208
- [Background] Chappell MC. Nonclassical renin-angiotensin system and renal function. Compr Physiol. 2012 Oct;2(4):2733-52. doi: 10.1002/cphy.c120002. PMID 23720263
- [Background] Bryniarski P, Nazimek K, Marcinkiewicz J. Immunomodulatory Activity of the Most Commonly Used Antihypertensive Drugs-Angiotensin Converting Enzyme Inhibitors and Angiotensin II Receptor Blockers. Int J Mol Sci. 2022 Feb 4;23(3):1772. doi: 10.3390/ijms23031772. PMID 35163696
- [Background] Persson PB. Renin: origin, secretion and synthesis. J Physiol. 2003 Nov 1;552(Pt 3):667-71. doi: 10.1113/jphysiol.2003.049890. Epub 2003 Aug 29. PMID 12949225
- [Background] Kotani Y, Belletti A, Maiucci G, Lodovici M, Fresilli S, Landoni G, Bellomo R, Zarbock A. Renin as a Prognostic Marker in Intensive Care and Perioperative Settings: A Scoping Review. Anesth Analg. 2024 May 1;138(5):929-936. doi: 10.1213/ANE.0000000000006682. Epub 2023 Oct 24. PMID 38358109
- [Background] Khanna AK. Tissue Perfusion and Prognosis in the Critically Ill-Is Renin the New Lactate? Crit Care Med. 2019 Feb;47(2):288-290. doi: 10.1097/CCM.0000000000003582. No abstract available. PMID 30653057
- [Background] See EJ, Chaba A, Spano S, Maeda A, Clapham C, Burrell LM, Liu J, Khasin M, Liskaser G, Eastwood G, Bellomo R. Renin Levels and Angiotensin II Responsiveness in Vasopressor-Dependent Hypotension. Crit Care Med. 2024 Aug 1;52(8):1218-1227. doi: 10.1097/CCM.0000000000006273. Epub 2024 Mar 21. PMID 38511994
- [Result] Qadri F, Culman J, Veltmar A, Maas K, Rascher W, Unger T. Angiotensin II-induced vasopressin release is mediated through alpha-1 adrenoceptors and angiotensin II AT1 receptors in the supraoptic nucleus. J Pharmacol Exp Ther. 1993 Nov;267(2):567-74. PMID 8246129
- [Result] Bellomo R, Wunderink RG, Szerlip H, English SW, Busse LW, Deane AM, Khanna AK, McCurdy MT, Ostermann M, Young PJ, Handisides DR, Chawla LS, Tidmarsh GF, Albertson TE. Angiotensin I and angiotensin II concentrations and their ratio in catecholamine-resistant vasodilatory shock. Crit Care. 2020 Feb 6;24(1):43. doi: 10.1186/s13054-020-2733-x. PMID 32028998
- [Result] Zhang W, Chen X, Huang L, Lu N, Zhou L, Wu G, Chen Y. Severe sepsis: Low expression of the renin-angiotensin system is associated with poor prognosis. Exp Ther Med. 2014 May;7(5):1342-1348. doi: 10.3892/etm.2014.1566. Epub 2014 Feb 20. PMID 24940436
- [Result] Bellomo R, Forni LG, Busse LW, McCurdy MT, Ham KR, Boldt DW, Hastbacka J, Khanna AK, Albertson TE, Tumlin J, Storey K, Handisides D, Tidmarsh GF, Chawla LS, Ostermann M. Renin and Survival in Patients Given Angiotensin II for Catecholamine-Resistant Vasodilatory Shock. A Clinical Trial. Am J Respir Crit Care Med. 2020 Nov 1;202(9):1253-1261. doi: 10.1164/rccm.201911-2172OC. PMID 32609011
- [Result] Prondzinsky R, Knupfer A, Loppnow H, Redling F, Lehmann DW, Stabenow I, Witthaut R, Unverzagt S, Radke J, Zerkowski HR, Werdan K. Surgical trauma affects the proinflammatory status after cardiac surgery to a higher degree than cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2005 Apr;129(4):760-6. doi: 10.1016/j.jtcvs.2004.07.052. PMID 15821641
- [Result] Hickey E, Karamlou T, You J, Ungerleider RM. Effects of circuit miniaturization in reducing inflammatory response to infant cardiopulmonary bypass by elimination of allogeneic blood products. Ann Thorac Surg. 2006 Jun;81(6):S2367-72. doi: 10.1016/j.athoracsur.2006.02.071. PMID 16731105
- [Result] Leisman DE, Fernandes TD, Bijol V, Abraham MN, Lehman JR, Taylor MD, Capone C, Yaipan O, Bellomo R, Deutschman CS. Impaired angiotensin II type 1 receptor signaling contributes to sepsis-induced acute kidney injury. Kidney Int. 2021 Jan;99(1):148-160. doi: 10.1016/j.kint.2020.07.047. Epub 2020 Aug 31. PMID 32882263
- [Result] Garcia B, Su F, Dewachter L, Favory R, Khaldi A, Moiroux-Sahraoui A, Annoni F, Vasques-Novoa F, Rocha-Oliveira E, Roncon-Albuquerque R Jr, Hubesch G, Njimi H, Vincent JL, Taccone FS, Creteur J, Herpain A. Myocardial effects of angiotensin II compared to norepinephrine in an animal model of septic shock. Crit Care. 2022 Sep 18;26(1):281. doi: 10.1186/s13054-022-04161-3. PMID 36117167
- [Result] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Result] Tumlin JA, Murugan R, Deane AM, Ostermann M, Busse LW, Ham KR, Kashani K, Szerlip HM, Prowle JR, Bihorac A, Finkel KW, Zarbock A, Forni LG, Lynch SJ, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Bellomo R; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Outcomes in Patients with Vasodilatory Shock and Renal Replacement Therapy Treated with Intravenous Angiotensin II. Crit Care Med. 2018 Jun;46(6):949-957. doi: 10.1097/CCM.0000000000003092. PMID 29509568
- [Result] Chawla LS, Busse L, Brasha-Mitchell E, Davison D, Honiq J, Alotaibi Z, Seneff MG. Intravenous angiotensin II for the treatment of high-output shock (ATHOS trial): a pilot study. Crit Care. 2014 Oct 6;18(5):534. doi: 10.1186/s13054-014-0534-9. PMID 25286986
- [Result] Wieruszewski PM, Bellomo R, Busse LW, Ham KR, Zarbock A, Khanna AK, Deane AM, Ostermann M, Wunderink RG, Boldt DW, Kroll S, Greenfeld CR, Hodges T, Chow JH; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Initiating angiotensin II at lower vasopressor doses in vasodilatory shock: an exploratory post-hoc analysis of the ATHOS-3 clinical trial. Crit Care. 2023 May 5;27(1):175. doi: 10.1186/s13054-023-04446-1. PMID 37147690
- [Result] Smith SE, Newsome AS, Guo Y, Hecht J, McCurdy MT, Mazzeffi MA, Chow JH, Kethireddy S. A Multicenter Observational Cohort Study of Angiotensin II in Shock. J Intensive Care Med. 2022 Jan;37(1):75-82. doi: 10.1177/0885066620972943. Epub 2020 Nov 24. PMID 33231111
- [Result] See EJ, Clapham C, Liu J, Khasin M, Liskaser G, Chan JW, Serpa Neto A, Costa Pinto R, Bellomo R. A PILOT STUDY OF ANGIOTENSIN II AS PRIMARY VASOPRESSOR IN CRITICALLY ILL ADULTS WITH VASODILATORY HYPOTENSION: THE ARAMIS STUDY. Shock. 2023 May 1;59(5):691-696. doi: 10.1097/SHK.0000000000002109. Epub 2023 Mar 18. PMID 36930693
- [Result] Wieruszewski PM, Wittwer ED, Kashani KB, Brown DR, Butler SO, Clark AM, Cooper CJ, Davison DL, Gajic O, Gunnerson KJ, Tendler R, Mara KC, Barreto EF. Angiotensin II Infusion for Shock: A Multicenter Study of Postmarketing Use. Chest. 2021 Feb;159(2):596-605. doi: 10.1016/j.chest.2020.08.2074. Epub 2020 Aug 31. PMID 32882250
- [Result] Coulson TG, Miles LF, Serpa Neto A, Pilcher D, Weinberg L, Landoni G, Zarbock A, Bellomo R. A double-blind randomised feasibility trial of angiotensin-2 in cardiac surgery. Anaesthesia. 2022 Sep;77(9):999-1009. doi: 10.1111/anae.15802. PMID 35915923
- [Result] Coulson TG, Miles LF, Zarbock A, Burrell LM, Patel SK, von Groote T, Pilcher D, Weinberg L, Landoni G, Bellomo R. Renin-angiotensin-aldosterone system dynamics after targeted blood pressure control using angiotensin II or norepinephrine in cardiac surgery: mechanistic randomised controlled trial. Br J Anaesth. 2023 Oct;131(4):664-672. doi: 10.1016/j.bja.2023.06.056. Epub 2023 Jul 20. PMID 37481435
- [Result] Wieruszewski PM, Seelhammer TG, Barreto EF, Busse LW, Chow JH, Davison DL, Gaglani B, Khanna AK, Ten Lohuis CC, Mara KC, Wittwer ED. Angiotensin II for Vasodilatory Hypotension in Patients Requiring Mechanical Circulatory Support. J Intensive Care Med. 2023 May;38(5):464-471. doi: 10.1177/08850666221145864. Epub 2022 Dec 15. PMID 36524274
- [Result] Wan L, Langenberg C, Bellomo R, May CN. Angiotensin II in experimental hyperdynamic sepsis. Crit Care. 2009;13(6):R190. doi: 10.1186/cc8185. Epub 2009 Nov 30. PMID 19948019
- [Result] Lankadeva YR, Kosaka J, Evans RG, Bellomo R, May CN. Urinary Oxygenation as a Surrogate Measure of Medullary Oxygenation During Angiotensin II Therapy in Septic Acute Kidney Injury. Crit Care Med. 2018 Jan;46(1):e41-e48. doi: 10.1097/CCM.0000000000002797. PMID 29077618
- [Result] Stolk RF, van der Pasch E, Naumann F, Schouwstra J, Bressers S, van Herwaarden AE, Gerretsen J, Schambergen R, Ruth MM, van der Hoeven JG, van Leeuwen H, Pickkers P, Kox M. Norepinephrine Dysregulates the Immune Response and Compromises Host Defense during Sepsis. Am J Respir Crit Care Med. 2020 Sep 15;202(6):830-842. doi: 10.1164/rccm.202002-0339OC. PMID 32520577
- [Result] Gleeson PJ, Crippa IA, Mongkolpun W, Cavicchi FZ, Van Meerhaeghe T, Brimioulle S, Taccone FS, Vincent JL, Creteur J. Renin as a Marker of Tissue-Perfusion and Prognosis in Critically Ill Patients. Crit Care Med. 2019 Feb;47(2):152-158. doi: 10.1097/CCM.0000000000003544. PMID 30653055
- [Result] Jeyaraju M, McCurdy MT, Levine AR, Devarajan P, Mazzeffi MA, Mullins KE, Reif M, Yim DN, Parrino C, Lankford AS, Chow JH. Renin Kinetics Are Superior to Lactate Kinetics for Predicting In-Hospital Mortality in Hypotensive Critically Ill Patients. Crit Care Med. 2022 Jan 1;50(1):50-60. doi: 10.1097/CCM.0000000000005143. PMID 34166293
- [Result] Leisman DE, Handisides DR, Busse LW, Chappell MC, Chawla LS, Filbin MR, Goldberg MB, Ham KR, Khanna AK, Ostermann M, McCurdy MT, Adams CD, Hodges TN, Bellomo R; ATHOS-3 Investigators. ACE inhibitors and angiotensin receptor blockers differentially alter the response to angiotensin II treatment in vasodilatory shock. Crit Care. 2024 Apr 18;28(1):130. doi: 10.1186/s13054-024-04910-6. PMID 38637829
- [Result] Lesnik P, Lysenko L, Krzystek-Korpacka M, Woznica-Niesobska E, Mierzchala-Pasierb M, Janc J. Renin as a Marker of Tissue Perfusion, Septic Shock and Mortality in Septic Patients: A Prospective Observational Study. Int J Mol Sci. 2022 Aug 15;23(16):9133. doi: 10.3390/ijms23169133. PMID 36012398
- [Result] Chung KS, Song JH, Jung WJ, Kim YS, Kim SK, Chang J, Park MS. Implications of Plasma Renin Activity and Plasma Aldosterone Concentration in Critically Ill Patients with Septic Shock. Korean J Crit Care Med. 2017 May;32(2):142-153. doi: 10.4266/kjccm.2017.00094. Epub 2017 May 31. PMID 31723628
- [Result] Nguyen M, Denimal D, Dargent A, Guinot PG, Duvillard L, Quenot JP, Bouhemad B. Plasma Renin Concentration is Associated With Hemodynamic Deficiency and Adverse Renal Outcome in Septic Shock. Shock. 2019 Oct;52(4):e22-e30. doi: 10.1097/SHK.0000000000001285. PMID 30407370
- [Result] Stanski NL, Pode Shakked N, Zhang B, Cvijanovich NZ, Fitzgerald JC, Jain PN, Schwarz AJ, Nowak J, Weiss SL, Allen GL, Thomas NJ, Haileselassie B, Goldstein SL. Serum renin and prorenin concentrations predict severe persistent acute kidney injury and mortality in pediatric septic shock. Pediatr Nephrol. 2023 Sep;38(9):3099-3108. doi: 10.1007/s00467-023-05930-0. Epub 2023 Mar 20. PMID 36939916
- [Result] Flannery AH, Ortiz-Soriano V, Li X, Gianella FG, Toto RD, Moe OW, Devarajan P, Goldstein SL, Neyra JA. Serum renin and major adverse kidney events in critically ill patients: a multicenter prospective study. Crit Care. 2021 Aug 14;25(1):294. doi: 10.1186/s13054-021-03725-z. PMID 34391450
- [Result] Zelniker TA, Kaya Z, Gamerdinger E, Spaich S, Stiepak J, Giannitsis E, Katus HA, Preusch MR. Relationship between markers of inflammation and hemodynamic stress and death in patients with out-of-hospital cardiac arrest. Sci Rep. 2021 May 11;11(1):9954. doi: 10.1038/s41598-021-88474-3. PMID 33976254
- [Result] Meersch M, Weiss R, Massoth C, Kullmar M, Saadat-Gilani K, Busen M, Chawla L, Landoni G, Bellomo R, Gerss J, Zarbock A. The Association Between Angiotensin II and Renin Kinetics in Patients After Cardiac Surgery. Anesth Analg. 2022 May 1;134(5):1002-1009. doi: 10.1213/ANE.0000000000005953. PMID 35171852
- [Result] Kullmar M, Saadat-Gilani K, Weiss R, Massoth C, Lagan A, Cortes MN, Gerss J, Chawla LS, Fliser D, Meersch M, Zarbock A. Kinetic Changes of Plasma Renin Concentrations Predict Acute Kidney Injury in Cardiac Surgery Patients. Am J Respir Crit Care Med. 2021 May 1;203(9):1119-1126. doi: 10.1164/rccm.202005-2050OC. PMID 33320784
- [Result] Eleuteri D, Montini L, Cutuli SL, Rossi C, Alcaro F, Antonelli M. Renin-angiotensin system dysregulation in critically ill patients with acute respiratory distress syndrome due to COVID-19: a preliminary report. Crit Care. 2021 Mar 1;25(1):91. doi: 10.1186/s13054-021-03507-7. No abstract available. PMID 33648544